CLINICAL TRIAL: NCT05127525
Title: Randomized, Double-Masked, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of IRX-101 Versus 5% Povidone-Iodine as an Ocular Surface Sterilizer
Brief Title: EffiCacy, Safety and ToLErability of a Novel Ocular ANtiseptic for Ocular Use (CLEAN)
Acronym: CLEAN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Adverse event
Sponsor: iRenix Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRX-2021-001
Record Dates: First submitted 2021-10-19; First posted 2021-11-19 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Macular Edema; Branch Retinal Vein Occlusion; Glaucoma/Closed Angle Glaucoma
MeSH Terms: conditions — Retinal Vein Occlusion; Glaucoma, Angle-Closure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test Drug (Experimental): IRX-101 drops instilled prior to intravitreal injection
  Interventions: Drug: IRX-101
- Control (Active Comparator): Povidone-Iodine/Betadine drops instilled prior to intravitreal injection
  Interventions: Drug: Control

INTERVENTIONS:
Drug: IRX-101 — IRX-101 to prevent infectious endophthalmitis following intravitreal injection therapy (IVT)
  Other Names: Test Arm 1
  Arms: Test Drug
Drug: Control — Providone-Iodine Betadine to prevent infectious endophthalmitis following intravitreal injection therapy (IVT)
  Arms: Control

SUMMARY:
This is a randomized, double-masked, multicenter, study to evaluate the efficacy, safety, and tolerability of IRX-101 versus 5% povidone-iodine (PI) in subjects receiving intravitreal anti-VEGF injections. The study will be conducted in up to 30 centers in the United States (US).

DETAILED DESCRIPTION:
Intravitreal injection therapy (IVT) of anti-vascular endothelial growth factor (VEGF) agents has transformed the treatment landscape of several retinal diseases, including exudative (wet) macular degeneration, retinal vein occlusion, diabetic macular edema, and choroidal neovascularization. The most common adverse effects of IVT occur due to the side effects of Povidone-Iodine 5% (PI; brand name: Betadine® 5%; Alcon, Fort Worth, TX), the antiseptic placed on the ocular surface prior to each injection. PI is nearly universally used to prevent ocular infection (endophthalmitis). PI leads to marked corneal epithelial toxicity in humans,6, 7 resulting in debilitating side effects including decreased visual acuity and pain that can last more than 3 days post-IVT. Post-IVT pain is severe enough to require oral analgesics in up to 30% of patients and is a frequent cause of treatment discontinuation. Therefore, there is an unmet need in ophthalmology for a potent ocular antiseptic with a superior safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving informed consent
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, ≥ 18 years of age and receiving intravitreal anti-VEGF injections in one or both eyes

Exclusion Criteria:

1. Current or past diagnosis of endophthalmitis
2. Current diagnosis of uveitis
3. Current use of viscous lidocaine products for ocular anesthesia prior to IVT
4. Currently receiving intravitreal steroid injections
5. Concurrent participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of infectious endophthalmitis after topical use of IRX-101 combined with IVT | 2 hours post-injection
  To evaluate the rate of infectious endophthalmitis after topical use of IRX-101 following intravitreal injection therapy (IVT) (% occurrence or rate of population randomized to IRX-101 test arm)

SECONDARY OUTCOMES:
Telephone questionnaire regarding patient-reported post-injection pain | 2 hours post-injection
  Telephone questionnaire with questions asked of patients regarding patient-reported post-injection pain compared to Providone-Iodine Betadine control group (three questions asked scale of 0 to 10, 0 being no pain to 10 being worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Smith, MD, MS, Study Chair — iRenix Medical
Locations (1):
- Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No